CLINICAL TRIAL: NCT03214341
Title: Assessment of Mediastinal Masses With Diffusion Weighted MR Imaging
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehad Mohammed Safwat Ali, Principal Investigator, Assiut University
Other Study IDs: MRIML
Record Dates: First submitted 2017-06-24; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Mediastinal Tumor
Keywords: mediastinal masses; MRI diffusion
MeSH Terms: conditions — Mediastinal Neoplasms | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: MRI diffusion — using MRI diffusion to differentiate between benign and malignant mediastinal masses

SUMMARY:
Differentiation between benign and malignant mediastinal tumors as well as characterization and grading of malignancy which is essential for treatment planning as well as for prognosis

DETAILED DESCRIPTION:
Differentiation between benign and malignant mediastinal tumors as well as characterization and grading of malignancy is essential for treatment planning as well as for prognosis .

MRI presents valuable diagnostic information in assessing the mediastinum. In addition, special applications have been developed over recent years diffusion-weighted magnetic resonance imaging is one such technique The advent of echo-planar imaging technique has rendered diffusion weighted imaging of the abdomen and thoracic cavity possible .

Quantitative assessment of the mediastinal mass is possible by calculation of apparent diffusion co-efficient value ,which is related to the proportion of extracellular and intracellular component.

The apparent diffusion co-efficient is inversely correlated with tissue cellularity. It is lower in viable tumor tissue with densely packed diffusion-hindering obstacles than in tissue with less densely packed obstacles such as tumor necrosis and benign tissue .

ELIGIBILITY:
Inclusion Criteria:

* Any age groups
* diagnosis of mediastinal mass (by Multislice Computed Tomography).

Exclusion Criteria:

* chemotherapy radiotherapy.
* thoracic surgery.
* cystic mass .
* mass with large amount of necrosis or calcification.
* contraindication of MRI (e.g. pacemakers , claustrophobia).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with mediastinal masses
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity of magnetic resonance imaging diffusion in mediastinal masses | up to one month

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Thabet Hussein, professor, Principal Investigator — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Differentiation between benign and malignant mediastinal tumors as well as characterization and grading of malignancy which is essential for treatment planning as well as for prognosis

REFERENCES:
- See also: the investigator had gained some information from this site — https://www.google.com.eg/url?sa=t&rct=j&q=&esrc=s&source=web&cd=2&cad=rja&uact=8&ved=0ahUKEwjuiIL17bHUAhXJIlAKHcKpBKgQFgguMAE&url=http%3A%2F%2Fwww.sciencedirect.com%2Fscience%2Farticle%2Fpii%2FS0378603X15002600&usg=AFQjCNEOdfnMGP4KT6xObmi_TubWRSJq4Q-